CLINICAL TRIAL: NCT01419769
Title: A Prospective, Multi-center, Non-blinded, Single-arm (Nonrandomized) Study of the AXIOS Stent and Delivery System
Brief Title: AXIOS Stent & Delivery System Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xlumena, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD00744
Record Dates: First submitted 2011-08-15; First posted 2011-08-18 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Pancreatic Pseudocyst(s)
Keywords: symptomatic pancreatic pseudocyst; pancreatic pseudocyst; transluminal drainage; minimally invasive; Nitinol stent; transmural endoscopic drainage; catheter based
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AXIOS Stent and Delivery System (Experimental)
  Interventions: Device: AXIOS Stent & Delivery System

INTERVENTIONS:
Device: AXIOS Stent & Delivery System — The AXIOS Stent & Delivery System study is a prospective, multi-center, non-blinded, single-arm(nonrandomized) study that will be conducted at up to 10 sites in the United States, European Community and/or Japan will enroll a total of 24 patients. A majority of the patients will be enrolled in the United States.
  Patients between the age of 18 and 75 scheduled for endoscopic drainage of symptomatic pancreatic pseudocysts that are equal or greater than 6 cm in diameter, adherent to the bowel wall, and have ≥ 70% fluid contents are potential study candidates.
  Study patients will undergo the following clinical follow-up evaluations of study endpoints conducted at 30 days, 60 days, 1 week post stent removal and possibly at 3 and 6 months post stent removal.

SUMMARY:
The Xlumena AXIOS Stent and Delivery System is an investigational device in the USA, and this study is being conducted under an Investigational Device Exemption (IDE) granted by the US Food and Drug Administration (FDA).

The study design is prospective, multi-center, non-blinded, single-arm (nonrandomized) study. Up to 10 sites in the United States, European Community and/or Japan will enroll a total of 24 patients. A majority of the patients will be enrolled in the United States.

Patients will be followed at (approximately) 30 days and/or 60 days depending upon pseudocyst resolution confirmation, at 1-week post-stent removal,and possibly at 3 and 6 month post-stent removal.

DETAILED DESCRIPTION:
OBJECTIVE:

To demonstrate the safety and effectiveness of the Xlumena AXIOS Stent and Delivery System for endoscopic drainage of pancreatic pseudocysts in patients with symptomatic pancreatic pseudocysts that are greater than or equal to 6 cm (≥6cm) in diameter, have ≥ 70% fluid contents and are adherent to the bowel wall.

STUDY DESIGN:

Prospective, multi-center, non-blinded, single-arm (nonrandomized) study

KEY ENDPOINTS:

Safety: The safety endpoint is freedom from major complications through the duration of the 1-week post-stent removal study period, defined as:

1. Access site-related bleeding requiring transfusion;
2. Access site-related infection requiring intravenous or intramuscular antibiotics and/or extended hospitalization;
3. Surgery for access-site related perforation;
4. Stent migration/dislodgement into the pseudocyst or enteral lumen;
5. Tissue injury, defined as ulceration to the submucosa at site of stent implant as observed to persist through 1-week post-stent removal.
6. Serious adverse event classified as implant-associated or implant/endoscopic procedure-associated;

Effectiveness:

1. Stent lumen patency at 30 days and/or 60 days
2. Stent removability at 30 days and/ or 60 days.
3. Technical success, defined as: placement of the AXIOS stent using the AXIOS delivery system and removal of the AXIOS stent using a standard endoscopic snare.
4. Clinical success, defined as: at least a 50% decrease in pseudocyst size, based on radiographic analysis, at 30 days and/or 60 days.

PATIENT POPULATION:

Patients between 18 and 75 years of age, suitable for transluminal drainage of symptomatic pancreatic pseudocysts that are greater than or equal to 6 cm in diameter and adherent to the bowel wall are candidates for study treatment.

FOLLOW-UP SCHEDULE:

Clinical follow-up evaluations of study endpoints will be conducted at 30 days and/or 60 days, 1 week post stent removal and possibly at 3 and 6 months post stent removal.

PLANNED NUMBER OF PATIENTS, SITES & REGIONS:

The target enrollment for the study is 24 subjects. Study will be conducted at up to 10 investigational sites in the United States, Japan and/or the European Community. A majority of the patients will be enrolled in the United States.

ELIGIBILITY:
Inclusion Criteria:

* (patients must meet all criteria)

  1. Age between 18 and 75 years old, male or female.
  2. Eligible for endoscopic intervention.
  3. Acceptable candidate for endoscopic transluminal pancreatic pseudocyst drainage
  4. Symptomatic pancreatic pseudocyst having the following characteristics:

     * Greater than or equal to 6 cm in size (based upon the maximum crosssectional area in the CT scan),
     * Adherent to bowel wall, and
     * ≥70% fluid content
  5. Patient understands the study requirements and the treatment procedures and provides written Informed Consent using a form that has been approved by the local Institutional Review Board or Ethics Committee before any study-specific tests or procedures are performed.
  6. Patient is willing to comply with all specified follow-up evaluations, including willingness to undergo a pre/post CT imaging study.

Exclusion Criteria:

* (patients meeting any of the below criteria will be excluded from study)

  1. <18 or >75 years of age
  2. Pancreatic pseudocysts having the following characteristics:

     * Require nasocystic drainage,
     * < 69% fluid content
  3. The fluid collection to be drained is an immature pseudocyst
  4. The fluid collection to be drained is a cystic neoplasm
  5. The fluid collection to be drained is a pseudoaneurysm
  6. The fluid collection to be drained is a duplication cyst
  7. The fluid collection to be drained is a non-inflammatory fluid collection
  8. There is more than one pseudocyst requiring drainage
  9. Abnormal coagulation:

     * INR > 1.5 and not correctable
     * presence of a bleeding disorder
     * platelets < 50,000/mm3
  10. Altered anatomy that precludes the physician's ability to deliver the stent (decision on a case by case basis).
  11. Intervening gastric varices or vessels within a one centimeter radius of the needle (visible using endoscopy or endoscopic ultrasound)
  12. Any prior true anaphylactic reaction to contrast agents, nitinol (nickel titanium), silicone or any other materials contacting the patient.
  13. Female of childbearing potential with a positive pregnancy test prior to the procedure or intends to become pregnant during the study.
  14. Currently participating in another investigational drug of device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - California Pacific Medical Center (CPMC), San Francisco, California
  - Unversity of Colorado Denver, Aurora, Colorado
  - Borland-Groover Clinic, Jacksonville, Florida
  - University of Chicago Medical Center (UCMC), Chicago, Illinois
  - Cornell University, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
- Hospital Costa del Sol, Marbella, Spain

REFERENCES:
- [Derived] Shah RJ, Shah JN, Waxman I, Kowalski TE, Sanchez-Yague A, Nieto J, Brauer BC, Gaidhane M, Kahaleh M. Safety and efficacy of endoscopic ultrasound-guided drainage of pancreatic fluid collections with lumen-apposing covered self-expanding metal stents. Clin Gastroenterol Hepatol. 2015 Apr;13(4):747-52. doi: 10.1016/j.cgh.2014.09.047. Epub 2014 Oct 5. PMID 25290534
- See also: click here for more information about the Sponsor — http://www.xlumena.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AXIOS Stent and Delivery System
Started | 33
Completed | 29
Not Completed | 4
Not completed — Did not receive the AXIOS stent | 3
Not completed — Not evaluable due to pigtail stents | 1

BASELINE CHARACTERISTICS:
Population: Patients between 18 and 75 years of age, suitable for transluminal drainage of symptomatic pancreatic pseudocysts that are greater than or equal to 6 cm in diameter and adherent to the bowel wall are candidates for study treatment.
Arm/Group | AXIOS Stent and Delivery System
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.6 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 30
  Spain | 3
Height [Mean (Standard Deviation); unit: inches] | 67.4 (3.9)
Weight [Mean (Standard Deviation); unit: pounds] | 169.5 (43.5)

OUTCOME MEASURES:

1. Primary Outcome: Safety - Freedom From Major Complications: Access Site-related Bleeding
Description: Subjects are free of access site-related bleeding requiring transfusion
Time Frame: Through the duration of the 1-week post-stent removal study period
Population: Intent-to-Treat population
Measure: Number; unit: percentage of patients
Arm/Group | AXIOS Stent and Delivery System
Number analyzed (Participants) | 33
percentage of patients | 100

2. Secondary Outcome: Effectiveness: Stent Lumen Patency at 30 Days and/or 60 Days
Description: Stent lumen patency at 30 days and/or 60 days.
Time Frame: Up to 60 days
Population: Patients treated per protocol with successful stent placement.
Measure: Number; unit: percentage of patients
Arm/Group | AXIOS Stent and Delivery System
Number analyzed (Participants) | 29
percentage of patients | 93.1

3. Secondary Outcome: Effectiveness: Stent Removability at 30 Days and/or 60 Days
Description: AXIOS stent removal was indicated at the time of pseudocyst resolution (≤ 3 cm diameter) or at 60 the day post procedure visit. Scheduled examination for pseudocyst resolution was designated at 30 days for removal if the pseudocyst resolution criterion was met. Otherwise, the stent was left in place for removal at the 60 day visit.
Time Frame: Up to 60 days
Population: Patients who had AXIOS stent successfully placed during index procedure.
Measure: Number; unit: percentage of patients
Arm/Group | AXIOS Stent and Delivery System
Number analyzed (Participants) | 30
percentage of patients | 96.7

4. Secondary Outcome: Effectiveness: Technical Success
Description: Placement of the AXIOS Stent using the AXIOS Delivery System and removal of the AXIOS Stent using a standard endoscopic snare.
Time Frame: Up to 60 days
Population: Intent-to-Treat population
Measure: Number; unit: participants
Arm/Group | AXIOS Stent and Delivery System
Number analyzed (Participants) | 33
participants
  Placement of AXIOS stent | 30
  Removal of AXIOS stent using standard endosc snare | 29

5. Secondary Outcome: Clinical Success
Description: Clinical success is defined as at least a 50% decrease in pseudocyst size, based on radiographic analysis, at 30 days and/or 60 days.
Time Frame: Up to 60 days
Population: Patients treated per protocol.
Measure: Number; unit: percentage of patients
Arm/Group | AXIOS Stent and Delivery System
Number analyzed (Participants) | 29
percentage of patients | 86.2

6. Primary Outcome: Safety - Freedom From Major Complications: Access Site-related Infection
Description: Subjects are free of access site-related infection requiring intravenous or intramuscular antibiotics and/or extended hospitalization
Time Frame: Through the duration of the 1-week post-stent removal study period
Population: Per protocol population
Measure: Number; unit: percentage of patients
Arm/Group | AXIOS Stent and Delivery System
Number analyzed (Participants) | 29
percentage of patients | 96.6

7. Primary Outcome: Safety - Freedom From Major Complications: Perforation
Description: Subjects are free of surgery for access-site related perforation
Time Frame: Through the duration of the 1-week post-stent removal study period
Population: Intent-to-Treat population
Measure: Number; unit: percentage of patients
Arm/Group | AXIOS Stent and Delivery System
Number analyzed (Participants) | 33
percentage of patients | 100

8. Primary Outcome: Safety - Freedom From Major Complications: Stent Migration/Dislodement
Description: Treated subjects are free of stent migration/ dislodgement into the pseudocyst or enteral lumen
Time Frame: Through the duration of the 1-week post-stent removal study period
Population: Per protocol population of subjects with stent successfully placed
Measure: Number; unit: percentage of patients
Arm/Group | AXIOS Stent and Delivery System
Number analyzed (Participants) | 29
percentage of patients | 96.6

9. Primary Outcome: Safety - Freedom From Major Complications: Tissue Injury
Description: Subjects are free of tissue injury (ulceration to the submucosa) at stent site persisting through 1-week post-stent removal.
Time Frame: Through the duration of the 1-week post-stent removal study period
Population: Per protocol population
Measure: Number; unit: percentage of patients
Arm/Group | AXIOS Stent and Delivery System
Number analyzed (Participants) | 29
percentage of patients | 100

10. Primary Outcome: Safety - Freedom From Major Complications: SAE's
Description: Treated subjects are free of serious adverse event classified as implant-associated or implant/endoscopic procedure-associated.
Time Frame: Through the duration of the 1-week post-stent removal study period
Population: Intent-to-Treat population
Measure: Number; unit: percentage of patients
Arm/Group | AXIOS Stent and Delivery System
Number analyzed (Participants) | 33
percentage of patients | 84.8

ADVERSE EVENTS:
Time Frame: From index procedure up to 6 months post-stent removal
Description: Events are categorized as Post-index Procedure, Early Post-Stent Removal (within 7 days of stent removal), and Late Post-Stent Removal (beyond 7 days)
Arm/Group | AXIOS Stent and Delivery System
Serious Adverse Events (participants affected / at risk) | 16/33
Other Adverse Events (participants affected / at risk) | 15/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXIOS Stent and Delivery System (N=33)
Abdominal Pain (Gastrointestinal disorders) | 6 (6)
Abdominal pain and nausea after eating (Gastrointestinal disorders) | 1 (1)
Abdominal pain and vomiting after eating (Gastrointestinal disorders) | 1 (1)
Abdominal pain, nausea, and vomiting after eating (Gastrointestinal disorders) | 1 (1)
Abdominal pain and syncope, GI bleeding (Gastrointestinal disorders) | 1 (1)
Nausea and vomiting only after eating (Gastrointestinal disorders) | 2 (2)
Infection (Infections and infestations) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Chest pain (Cardiac disorders) | 1 (1)
Chest pain and pressure, shortness of breath, heart palpitations (Cardiac disorders) | 1 (1)
Fever (Infections and infestations) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 1 (1)
Headache and lightheadedness/ dizziness (Nervous system disorders) | 1 (1)
Intraperitoneal air (Gastrointestinal disorders) | 1 (1)
Left shoulder/ back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Respiratory failure (Cardiac disorders) | 1 (1)
Severe dehydration (General disorders) | 1 (1)
Mucus overgrowth (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXIOS Stent and Delivery System (N=33)
Abdominal Pain (Gastrointestinal disorders) | 9 (11)
Nausea after eating (Gastrointestinal disorders) | 5 (5)
Fever (Infections and infestations) | 4 (4)
Vomiting after eating (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Lightheadedness/ dizziness (General disorders) | 2 (2)
New pancreatic pseudocyst (Gastrointestinal disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Black stool (Gastrointestinal disorders) | 1 (1)
Bleeding (General disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flank pain (General disorders) | 1 (1)
J-tube clogged (Gastrointestinal disorders) | 1 (1)
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic duct obstruction (Gastrointestinal disorders) | 1 (1)
Peripancreatic inflammation (Gastrointestinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must wait 9 months after close of study for Sponsor to present collaborative publication. If Sponsor does not publish within 9 months after close of study, PI is free to publish institution's results at that time.

Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of 6 months from the date the PI receives the objection. The Sponsor cannot require changes to the communication and cannot extend the embargo.